CLINICAL TRIAL: NCT01573026
Title: Clinical Analysis of a Biomimetic Implant System: Five Year Survival Rates, Marginal Bone-level Changes, and Soft Tissue Aesthetics.
Brief Title: Five Year Survival Study Evaluating the Genesis Dental Implant System
Acronym: Genesis Dental
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Keystone Dental, Inc. (Industry)
Collaborators: Aptiv Solutions (Industry); Pirkka Nummikoski, DDS, MS (Unknown); CadBlu North (Hastings, MN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: KD-CR 02
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Dental Implants
Keywords: Dental Implants; Dental Implantation; Osseointegration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to document the use if the Keystone Dental Genesis Dental Implant System in standard clinical use and to provide 5 year survival data.

DETAILED DESCRIPTION:
The technology behind dental implants is well established and the Genesis Dental Implant System has been cleared for marketing by the FDA. It is Keystone Dental's choice to collect post-market data within the framework of a clinical trial in order to assess the clinical performance of this device.

The risks of the Genesis Dental Implant System are no different than other comparable dental implant systems currently in use. Keystone Dental expects the clinical performance of this device to be equal to that of comparable implant systems.

The purpose of this research study is to assess the 5 year survival rate of the Genesis Dental Implant System, as well as assess the safety and effectiveness endpoints, which include incidence of adverse effects, change in bone height and soft tissue aesthetic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 18 and 85 years old, inclusive, and have passed growth maximum at the time of implant placement
* Subject must be willing to sign the informed consent document and adhere to study procedures.
* Subject must have one or more natural teeth missing or about to be extracted.
* Subject must fulfill all the accepted medical and dental requirements for treatment with dental implants.
* Subject must desire treatment with dental implants.

Exclusion Criteria:

* Subject refuses to sign the informed consent document.
* Subject's treatment success by both clinical and esthetic measures may be compromised by the restricted range of product available for the study.
* The treatment plan to use the range of products available is not in the best interests of the subject. Please see Section 1.2.1 for restrictions on product availability.
* The implant site(s) had a previously failed implant.
* Subject cannot be treated within the restrictions of the treatment plan laid out in Section 5. In addition, please see Section 1.2.1 for restrictions on product availability.
* Subject with alveolar ridge dimensions that are not sufficient to accommodate and sustain proper implant placement.
* Subject is not communicable in an understandable language.
* Current Alcohol or Drug Abuse (within previous 12 months) as noted in the subject's chart.
* Women who are pregnant at time of enrollment in to the study.
* Subject with out of control metabolic disease.
* Subject who have been on chemotherapy or long term cortisone use (at any time).
* Subject with known allergy to titanium.
* Subject with diabetes.
* Subject with a history of autoimmune disease (e.g. documented multiple allergies, systemic lupus erythematosus, dermatomyositis, etc.) or immunosuppressive disease (e.g. human immunodeficiency virus or acquired immunodeficiency syndrome).
* Subject with epilepsy.
* Subjects with uncontrolled or severe cases of hyperthyroidism, malignancies, renal disease, liver problems, hypertension, leukemia, severe vascular heart disease, hepatitis, collagen and bone diseases, or other serious illnesses.
* Subject currently taking bisphosphonate or calcium channel blockers.
* There is reasonable doubt that the subject will comply with the recall schedule.
* There is reasonable doubt that the subject will comply with the clinicians' instructions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects between the ages of 18 and 85 who require dental implants
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Tarnow, DDS, Principal Investigator — Specialized Dentistry of New York
Locations (8):
- United States (8):
  - Newport Coast Oral Facial Institute, Newport Beach, California
  - Brighton Periodontal & Implant Dental Group, Woodland Hills, California
  - Periodontal Medicine & Surgical Specialists, LTD, Oakbrook Terrace, Illinois
  - Kevin G. Murphy & Associates, PA, Baltimore, Maryland
  - Specialized Dentistry of New York, New York, New York
  - Edwin Rosenberg, DMD, HDD, BDS, Philadelphia, Pennsylvania
  - PerioHealth Professionals, PLLC, Houston, Texas
  - Dental Design, Gainesville, Virginia